CLINICAL TRIAL: NCT04247906
Title: Single Patient Expanded Access Treatment Plan (EAP; Also Known As A Compassionate Use Plan) To Provide Patients Access To The Investigational Product Narsoplimab
Brief Title: Single Patient Expanded Access Treatment Plan For The Investigational Product Narsoplimab
Status: Available | Type: Expanded Access
Sponsor: Omeros Corporation (Industry)
Collaborators: Impatients N.V. trading as myTomorrows (Industry)
Responsible Party: Sponsor
Other Study IDs: 721-TMA-EA
Record Dates: First submitted 2020-01-28; First posted 2020-01-30 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Hematopoietic Stem Cell Transplant Associated Thrombotic Microangiopathy (HSCT-TMA)
MeSH Terms: interventions — narsoplimab

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: Narsoplimab
  Other Names: OMS721

SUMMARY:
The purpose of the EAP is to provide access to hematopoietic stem cell transplant-associated thrombotic microangiopathy (HSCT-TMA) patients who may benefit from treatment with narsoplimab based on the medical judgement of their respective physicians.

ELIGIBILITY:
* Patient (adult or pediatric) must have undergone allogeneic or autologous hematopoietic stem cell transplant (HSCT)
* Patient must be capable of understanding an informed consent form (ICF) or the parent or legal guardian of the patient is able to understand and sign a written ICF prior to the initiation of any treatment procedures.
* Patient must have HSCT- TMA defined as having thrombocytopenia and evidence of microangiopathic hemolytic anemia.

Sex: All
Age Groups: Child, Adult, Older Adult